CLINICAL TRIAL: NCT06731478
Title: A Multicenter, Randomized, Open-Label, Phase 3 Trial of Trastuzumab Deruxtecan (Enhertu®) Plus Chemotherapy Plus or Minus Pembrolizumab Versus Chemotherapy Plus Trastuzumab Plus or Minus Pembrolizumab as First-Line Treatment in Participants With Unresectable, Locally Advanced or Metastatic HER2-Positive Gastric Or Gastroesophageal Junction (GEJ) Cancer (Destiny-Gastric05)
Brief Title: Study of TDXd, Chemotherapy, Pembrolizumab, and Trastuzumab in First-Line Metastatic HER2-Positive Gastric or Gastroesophageal Junction Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-724; KEYNOTE-G03 (Other: Merck Sharp & Dohme LLC); MK-3475-G03 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Enhertu; Trastuzumab Deruxtecan; Chemotherapy; DS-8201a; HER2 positive
MeSH Terms: conditions — Stomach Neoplasms | interventions — trastuzumab deruxtecan; pembrolizumab; Trastuzumab; Drug Therapy

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Main Cohort: Arm M1 (Experimental): Participants will receive T-DXd plus fluoropyrimidine (5-FU or capecitabine) plus pembrolizumab
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: pembrolizumab; Drug: Chemotherapy
- Main Cohort: Arm M2 (Experimental): Participants will receive Trastuzumab plus platinum-based chemotherapy (cisplatin plus 5-FU or oxaliplatin plus capecitabine) plus pembrolizumab
  Interventions: Drug: pembrolizumab; Drug: Trastuzumab; Drug: Chemotherapy
- Exploratory Cohort: Arm E1 (Experimental): Participants will receive T-DXd plus fluoropyrimidine (5-FU or capecitabine)
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: Chemotherapy
- Exploratory Cohort: Arm E2 (Experimental): Participants will receive Trastuzumab plus platinum-based chemotherapy (cisplatin plus 5-FU or oxaliplatin plus capecitabine)
  Interventions: Drug: Trastuzumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — T-DXd will be administered at a dose of 5.4 mg/kg intravenously (IV) every 3 weeks (Q3W)
  Other Names: T-DXd; ENHERTU®; DS-8201a
  Arms: Exploratory Cohort: Arm E1; Main Cohort: Arm M1
Drug: pembrolizumab — Pembrolizumab will be administered at a dose of 200 mg IV Q3W
  Other Names: KEYTRUDA®
  Arms: Main Cohort: Arm M1; Main Cohort: Arm M2
Drug: Trastuzumab — Trastuzumab will be administered at a loading dose of 8 mg/kg IV followed by 6 mg/kg IV Q3W
  Arms: Exploratory Cohort: Arm E2; Main Cohort: Arm M2
Drug: Chemotherapy — For Arms M1 and E1: 5-FU or capecitabine will be administered.
  For Arms M2 and E2: Cisplatin plus 5-FU or oxaliplatin plus capecitabine will administered.

SUMMARY:
This clinical trial is designed to assess the efficacy and safety of the triplet combination of trastuzumab deruxtecan (ENHERTU, T-DXd, DS-8201a) plus a fluoropyrimidine plus pembrolizumab versus standard of care (SoC) chemotherapy plus trastuzumab plus pembrolizumab as first-line therapy in participants with unresectable, locally advanced or metastatic HER2-positive tumor PD-L1 CPS ≥1 gastric or GEJ cancer in the Main Cohort. An Exploratory Cohort will also be evaluated to assess the efficacy and safety of T-DXd plus a fluoropyrimidine versus SoC chemotherapy plus trastuzumab in participants with unresectable, locally advanced or metastatic HER2-positive tumor PD-L1 CPS <1 gastric or GEJ cancer.

ELIGIBILITY:
Inclusion

1. Sign and date the Tissue Prescreening ICF, prior to HER2 and PD-L1 CPS central testing. Sign and date the Main Screening ICF, prior to the start of any trial-specific qualification procedures. Sign and date the Optional PGx ICF (included in the Main Screening ICF) prior to any PGx procedure.
2. Adults ≥18 years of age on the day of signing the ICF. Follow local regulatory requirements if the legal age of consent for trial participation is >18 years old.
3. Previously untreated, unresectable, locally advanced or metastatic gastric or GEJ adenocarcinoma histologically confirmed by pathology report. Prior treatment in the perioperative and/or adjuvant setting is permissible, provided there is >6 months between the end of perioperative or neoadjuvant treatment and the diagnosis of recurrent disease.

   Note: Prior use of IO (ie, anti-PD-1/PD-L1) therapy in the (neo)adjuvant setting is allowed as long as there is >6 months between the end of IO therapy and the diagnosis of recurrent disease.
4. Centrally determined HER2-positive (IHC 3+ or IHC 2+/ISH-positive) gastric or GEJ cancer as classified by the American Society of Clinical Oncology-College of American Pathologists for GC on a tumor biopsy as detected by prospective central test on new (core, incisional, excisional biopsy) or existing tumor tissue taken at the time of diagnosis of locally advanced or metastatic disease.

   Note: Archival samples taken from a previous diagnostic or surgical biopsy not previously irradiated can be accepted. Details pertaining to tumor tissue submission can be found in the Study Laboratory Manual.
5. All participants must provide a tumor sample for tissue-based IHC staining to centrally determine HER2 expression, PD-L1 CPS, and other correlatives. The mandatory FFPE tumor sample can be from either the primary tumor or metastatic biopsy. Specimens with limited tumor content (as centrally determined) and cytology samples are inadequate for defining tumor HER2 and PD-L1 status.
6. At least 1 target measurable lesion on CT or MRI, assessed by the investigator based on RECIST v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
7. LVEF ≥50% within 28 days before randomization.

exclusion criteria

1. Prior exposure to other HER2-targeting therapies (including ADCs).
2. Lack of physiological integrity of the upper gastrointestinal tract (ie, severe Crohn disease that results in malabsorption) or malabsorption syndrome that would preclude feasibility of oral chemotherapy (ie, capecitabine).
3. Known DPD enzyme deficiency. Note: Screening for DPD enzyme deficiency is required only in regions/countries where DPD testing is SoC and with unknown DPD status. For regions/countries where DPD testing is not SoC, local practice should be followed.
4. Contraindications to trastuzumab, 5-FU, capecitabine, cisplatin, or oxaliplatin treatment as per local label.
5. Medical history of myocardial infarction within 6 months before randomization or symptomatic CHF (New York Heart Association Class II to IV). Participants with troponin levels above ULN at Screening (as defined by the manufacturer) and without any myocardial infarction -related symptoms should have a cardiologic consultation during the Screening Period to rule out myocardial infarction.
6. Has a corrected QT interval (QTcF) prolongation to >470 ms (females) or >450 ms (males) based on the average of the screening triplicate 12-lead ECG.
7. Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening
8. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within 3 months of the trial randomization, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization to the date of radiographic disease progression or death due to any cause, up to 59 months
  PFS is defined as the time interval from the date of randomization to the date of radiographic disease progression as assessed by blinded independent central review (BICR) based on RECIST v1.1 or death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization to the date of death due to any cause, up to 59 months
  OS is defined as the time interval from the date of randomization to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (248):
- United States (18):
  - Yale Cancer Center, New Haven, Connecticut
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center - MAIN, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Prisma Health Cancer Institute, ITOR, CRU, Greenville, South Carolina
  - Tennessee Oncology Nashville Midtown, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Argentina (5):
  - CEMIC Ciudad Autonoma, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Clinica Universitaria Privada Reina Fabiola, Córdoba
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
- Australia (7):
  - Flinders Medical Centre, Bedford Park
  - Monash Medical Centre Clayton, Clayton
  - Townsville University Hospital, Douglas
  - Peter MacCallum Cancer Centre, North Melbourne
  - GenesisCare North Shore (Oncology), St Leonards
  - St John of God Subiaco Hospital, Subiaco
  - Wollongong Hospital, Wollongong
- Austria (5):
  - LKH - Universitaetsklinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
  - St. Josef Krankenhaus Wien, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (6):
  - Institut Jules Bordet, Anderlecht
  - AZ Sint-Lucas, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - CHU UCL Namur, Namur
- Brazil (12):
  - Centro de Oncologia - Unidade Brasilia - Hospital Sirio Libanes, Brasília
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira Sao Paulo, Brazil
  - CEPON - Centro de Pesquisas Oncológicas de Santa Catarina, Florianópolis
  - Fundação Doutor Amaral Carvalho, Jaú
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - IMIP - Instituto de Medicina Integral Professor Fernando Figueira, Recife
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - Obras Sociais Irmã Dulce - Hospital Santo Antônio, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, Sao Jose Rio Preto
- Canada (7):
  - Cité de la Santé de Laval, Laval
  - Trillium Health Partners Credit Valley Hospital, Mississauga
  - St. Mary's Hospital, Montreal
  - CHUS - Hôtel-Dieu, Sherbrooke
  - Mount Sinai Hospital, Toronto
  - Sunnybrook Health Sciences Centre, Toronto
  - University Health Network - Princess Margaret Cancer Centre, Toronto
- Chile (6):
  - Biocenter, Concepción
  - URUMED Spa, Rancagua
  - Centro de Investigacion del Maule, Region Del Maule
  - Centro de Estudios Clinicos SAGA, Santiago
  - FALP - Fundación Arturo López Pérez, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
- China (26):
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Fujian Cancer Hospital, Fuzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Zhejiang University school of medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Gansu Provincial Cancer Hospital, Lanzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Linyi Cancer Hospital, Linyi
  - Meizhou People's Hospital, Meizhou
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Shanxi Provincial People's Hospital, Taiyuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Affiliated Cancer Hospital of Xinjiang Medical university, Ürümqi
  - Hubei Cancer Hospital, Wuhan
  - Wuxi 4th People's Hospital, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Fudan University Shanghai Cancer Center, Xuhui District
  - Xuzhou Central Hospital, Xuzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
- France (16):
  - Institut Sainte Catherine, Avignon
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - Centre Georges François Leclerc, Dijon
  - CHU Grenoble - Hopital Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - Hopital Prive Jean Mermoz, Lyon
  - CHU Montpellier, Saint Eloi, Montpellier
  - Chru De Nantes Hotel-Dieu, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint-Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - Institut de Cancérologie de Strasbourg Europe - ICANS, Strasbourg
  - Hôpital Foch, Suresnes
  - Hopital Rangueil, Toulouse
- Germany (9):
  - Charité Universitätsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Klinikum rechts der Isar der TU Muenchen, München
- Italy (16):
  - Presidio Ospedaliero Garibaldi Nesima, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florenze
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Unità Sanitaria Locale- Ravenna, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Card. G. Panico, Tricase
- Japan (17):
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūōku
  - Gifu University Hospital, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa-shi
  - JCHO Kyushu Hospital, Kitakyushu
  - Kochi Health Sciences Center, Kochi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - NHO Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center Hospital, Nagoya
  - Miyagi Cancer Center, Natori-shi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osakasayama-shi
  - Hokkaido University Hospital, Sapporo
  - Osaka University Hospital, Suita-shi
  - Kanagawa Cancer Center, Yokohama
- Netherlands (6):
  - Antoni van Leeuwenhoek, Amsterdam
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - ETZ Elisabeth, Tilburg
  - UMC Utrecht, Utrecht
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Akershus universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Ullevål, Oslo
  - St. Olavs Hospital Hf, Universitetssykehuset i Trondheim, Trondheim
- Poland (5):
  - Beskidzkie Centrum Onkologii im.Jana Pawla II, Bielsko-Biala
  - Szpital Wojewodzki im. Mikolaja Kopernika, Koszalin
  - Wielkopolskie Centrum Onkologii, Poznan
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej Curie Panstwowy Instytut Badawczy W Warszawie, Warsaw
  - Warszawski Uniwersytet Medyczny, Warsaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimarães, E.P.E., Guimarães
  - Fundação Champalimaud, Lisbon
  - Hospital da Luz, Lisbon
  - Unidade Local de Saúde de Santa Maria, E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (7):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca
  - S.C Medisprof S.R.L, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie Craiova, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - S.C Ovidius Clinical Hospital S.R.L, Ovidiu
  - S.C. Sigmedical Services SRL, Suceava
- South Korea (14):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk national university hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (17):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Elche, Elche
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan
- Thailand (5):
  - Siriraj Hospital, Bangkoknoi
  - Vajira Hospital, Dusit
  - Songklanagarind Hospital, Hat Yai
  - Chulabhorn Hospital, Laksi
  - King Chulalongkorn Memorial Hospital, Pathum Wan
- Turkey (Türkiye) (10):
  - Medical Park Seyhan Hospital, Adana
  - Ankara City Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Dicle University, Medical faculty, Diyarbakır
  - Ataturk University Medical Faculty, Erzurum
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - İ.E.Ü. Medicalpoint İzmir Hastanesi, Izmir
  - Medical Park Samsun Hastanesi, Samsun
- United Kingdom (10):
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Cancer Centre, Cardiff
  - Ninewells Hospital, Dundee
  - Castle Hill Hospital, Hull
  - St James's University Hospital, Leeds
  - Sarah Cannon Research Institute UK, London
  - University College London Hospitals, London
  - Altnagelvin Area Hospital, Londonderry
  - The Christie Hospital, Manchester
  - Royal Marsden Hospital, Sutton
- Vietnam (5):
  - Hanoi Oncology hospital, Hanoi
  - National Cancer Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City
  - HCMC Oncology Hospital, Ho Chi Minh City
  - HCMC University Medical Center, HoChiMinh

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/